CLINICAL TRIAL: NCT07218770
Title: A Phase 1/2a Study of REGN7041 (Anti-CD3 Monoclonal Antibody) in Participants With Active Noninfectious Uveitis Affecting the Posterior Segment
Brief Title: A Study of REGN7041 for Active Noninfectious Uveitis in Adult Participants
Acronym: TITAN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R7041-NIU-24123; 2025-521713-57-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Active Noninfectious Uveitis Affecting the Posterior Segment
Keywords: NIU-PS; Intermediate; Posterior; Panuveitis; Anterior; Uveitis; Angiographic Cystoid Macular Edema (CME); Retinal vascular leakage
MeSH Terms: conditions — Panuveitis; Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequential Single Ascending Dose Cohorts (Experimental)
  Interventions: Drug: REGN7041
- Sequential Multiple Ascending Dose Cohorts (Experimental)
  Interventions: Drug: REGN7041

INTERVENTIONS:
Drug: REGN7041 — Administered as per the protocol

SUMMARY:
This study is researching an experimental drug called REGN7041 (also referred to as "study drug"). The study is focused on patients who have active inflammation inside of the eye without any signs of infection.

The aim of the study is to see how safe and tolerable the study drug is. This is the first time the study drug is being tested in humans.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood and the fluid in the eye at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of non-infectious anterior, intermediate, posterior or panuveitis (For anterior uveitis, there must be evidence of inflammation affecting the posterior segment), as defined in the protocol
2. Active disease at baseline, as defined in the protocol
3. Part A only: Best Corrected Visual Acuity (BCVA) of ≤65 and >10 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (Snellen equivalent of worse than or equal to 20/50 and better than 20/630) at the screening visit and on day 1
4. Part B only: BCVA of <75 and >10 ETDRS letters (Snellen equivalent of worse than 20/32 and better than 20/630) at the screening visit and on day 1

Key Exclusion Criteria:

1. BCVA of ≤30 ETDRS letters (Snellen equivalent of 20/250 or worse) at the screening visit and/or on day 1
2. Intraocular Pressure (IOP) <5 mm Hg at the screening visit and/or on day 1
3. IOP >25 mm Hg on day 1. Participants are permitted to take IOP-lowering eye drops
4. Confirmed or suspected infectious uveitis, as defined in the protocol

NOTE: Other Protocol-Defined Inclusion/Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2028-06-28 (Estimated); Study Completion 2028-06-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Through Week 24

SECONDARY OUTCOMES:
Concentrations of REGN7041 in serum | Through Week 24
Incidence of Anti-Drug Antibodies (ADAs) to REGN7041 in serum | Through Week 24
Magnitude of ADAs to REGN7041 in serum | Through Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Illinois Retina Associates, Oak Park, Illinois
  - Tennessee Retina PC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/